CLINICAL TRIAL: NCT03097185
Title: Analysis of Graft Function Following Autologous Islet Transplantation
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 010-150
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pancreatitis
Keywords: pancreatitis; islet cell
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each subject will provide samples of blood at specific timepoints as outlined in the protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analyze inflammatory markers and islet graft function through blood samples collected from subjects with chronic pancreatitis who undergo total pancreatectomy with auto islet transplantation.

DETAILED DESCRIPTION:
A total of 100 subjects will be enrolled in this study; 85 subjects will be enrolled from patients who are scheduled for TP-AIT and 15 subjects will be for TP alone at Baylor University Medical Center at Dallas or Baylor All Saints Medical Center at Fort Worth. The patients who are enrolled in a clinical study, named 'A phase 2/3, multicenter, randomized, double-blind, placebo-controlled, parallel assignment study to assess the efficacy and safety of reparixin in pancreatic islet auto-transplantation (REP0112, IND# 117390)', can be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic pancreatitis and who are scheduled for TP alone or TP-AIT
2. Patients aged 18 or older
3. Patients are able and willing to attend required follow-up visits at Baylor

Exclusion Criteria:

1. Patients who are unable/unwilling to attend follow-up visits at Baylor
2. For TP-AIT subjects: Patients who have advanced stage of chronic pancreatitis. The principal investigator or co-investigators carefully review the medical charts, laboratory results and radiology department reports and determine the suitability for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll a total of 100 patients for this study; 85 patients who will undergo with TP-AIT and 15 patients with TP alone.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-06-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of graft function following autologous islet transplantation | One year after transplant of islet cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E Beecherl, MD, Principal Investigator — Sammons Cancer Center, Baylor University Medical Center
Locations (1):
- Baylor University Medical Center - Sammons Outpatient Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided